CLINICAL TRIAL: NCT05243459
Title: Testing the Efficacy of an Eye-tracking-based Treatment in Reducing Stress-related Symptoms in Veterans With PTSD
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to the war that is taking place in Israel since October 7, 2023 and the high rates of active army reserve service among the population of the study.
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAU-GCFTveterans
Record Dates: First submitted 2022-01-27; First posted 2022-02-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gaze-Contingent Feedback Training (Experimental): In the task, 30 different matrices, each consisting of 16 faces, will be presented. Each matrix includes 8 angry faces and 8 neutral, 8 women and 8 men, and the locations are counterbalanced between matrices. The participants are asked to view the matrices in any way they choose, and the eye-tracking camera records their viewing location relative to the stimuli presented on the screen. At the beginning of each training session, the veteran will choose to which music he would like to listen during the 12-minute session from a diverse list of music. After calibrating the eye-tracking technology, the veteran will be instructed to view the matrices of faces as he chooses, as described above in the assessment task. The music chosen by the veteran will play only when s/he is looking at neutral faces and it will stop when s/he looks at threatening faces.
  Interventions: Behavioral: Gaze-Contingent Feedback Training
- RT-Based Attention Bias Modification (Active Comparator): The task consists of 160 trials. Each trial begins with a centrally-presented fixation cross (+), on which the participant is asked to focus for 500ms. When it disappears, two stimuli will be presented 1.5cm above and below the previous fixation cross for 500ms. After the stimuli disappear, a target probe (right- or left-pointing arrowhead) will appear in place of one of the stimuli, and the participant will be asked to indicate which target probe is presented by pressing the respective key. The target probe will remain on the screen until the participant's response, after which a new trial will begin.
  Participants are instructed to identify the probe type as quickly and accurately as possible.
  In the training task, all of the target probes will appear in the neutral face location. Thus, over multiple trials, learning occurs that the threatening face predicts the location of the target probe, thereby achieving the desiring change in attention patterns.
  Interventions: Behavioral: Attention Bias Modification
- Non-Contingent Feedback Training (Placebo Comparator): This condition is based on the aforementioned eye-tracking task with a fundamental change - The music chosen by the veteran will play continuously without any reinforcement for looking at threat or neutral faces.
  Interventions: Behavioral: Non-Contingent Feedback Training

INTERVENTIONS:
Behavioral: Gaze-Contingent Feedback Training — Feedback according to participants' viewing patterns, in order to modify their attention away from threat face stimuli.
  Arms: Gaze-Contingent Feedback Training
Behavioral: Attention Bias Modification — Attention training via repeated trials of a dot-probe task intended to direct attention away from threat stimuli using threat and neutral face stimuli.
  Arms: RT-Based Attention Bias Modification
Behavioral: Non-Contingent Feedback Training — Participants listen to a musical track they chose while viewing the face matrices. The music is played throughout and is not contingent upon gaze behavior.
  Arms: Non-Contingent Feedback Training

SUMMARY:
The study will examine the efficacy of a feedback-based treatment applying eye-tracking (Gaze-Contingent Music Reward Therapy) to change attention and gaze patterns associated with angry faces relative to a response-time-based attention bias modification treatment applying the dot-probe task and a control group.

DETAILED DESCRIPTION:
The study will recruit veterans with posttraumatic stress disorder (PTSD) due to a trauma acquired during military service. A compatibility check and initial filtering will happen via phone call, using basic symptom questionnaires for self-report and initial examination of exclusion criteria.

This study has four phases:

1. Clinical Assessment - Participants who pass the initial filtering and express a desire to participate in the study will be invited to a structured clinical interview during which clinical and practical inclusion and exclusion criteria will be examined by an independent evaluator (a clinical psychologist). After an explanation about the study and provision of signed informed consent from the participant, the clinical interview (CAPS-5 and MINI) will be conducted and self-report questionnaires will be completed:

   * Post-trauma Checklist (PCL) - PTSD symptoms
   * Patient Health Questionnaire (PHQ) - Depression Symptoms
   * Attention Bias Questionnaire (ABQ) - Attention Patterns
   * Attention Control Scale (ACS) - Attention Control
2. Attention bias measurement - participants will perform computerized tasks aimed to measure their attention bias prior to treatment.

   * Free viewing of 30 matrices each with 16 faces (8 with neutral facial expression and 8 with angry facial expression) while monitoring gaze location with passive eye-tracking technology - duration of this assessment is about 15 minutes.
   * Attention bias measurement using a dot-probe task in which two faces are presented on the screen and replaced by an arrow pointing right or left, and the participant has to indicate the arrow's direction by pressing a key - duration of the task is about 5 minutes.
   * Generic Flanker attention task, in which a middle arrow is presented with additional arrows to the right and left (for example <<><< or >>>>>) and the participant is asked to identify the direction of the middle arrow by pressing a key - duration of the task is about 5 minutes.
3. Attention Training - Next participants will be randomly assigned to one of three groups.

   * 8 sessions of Gaze Contingent Music Reward Therapy (GC-MRT) - In every session, the participant chooses music to which to listen and is then asked to view matrices of 16 faces as described above. The music plays when the participant views neutral faces and stops when viewing angry faces - each meeting lasts about 20 minutes.
   * 8 sessions of Attention Bias Modification Treatment based on a dot-probe task described above with one difference: While in the assessment task the probe location is counterbalanced at neutral and angry faces locations, in the treatment task the arrow always appears at the neutral face location - each session takes about 20 minutes.
   * Control group in which participants are exposed to the same procedure as GC-MRT but the music will play continually without contingency to participant's gaze.
4. Post-Training Assessment and Measurements - After the 8 treatment sessions, participants will undergo another clinical interview and the same questionnaires and attention assessment tasks similar to those conducted before the treatment. The clinical interview, questionnaires, and attention measurements will occur again after three months from the end of treatment (follow-up).

   * NOTE: As a direct result of the ongoing war in Israel the study has encountered serious difficulties in veteran-patients recruitment. First, many veterans were called into active duty since October 7th, 2023, limiting their availability for treatment/research. Second, with the war, numerous new treatment options have become available for veterans with PTSD, making it extremely difficult to recruit patients into a trial.

To date (March 18, 2025), 113 (target n=150) veterans have enrolled in the study and started treatment. Blinded group sizes from stratified randomization thus far stand at 39, 38, and 36.

Given this situation, we are forced to terminate the study early on June 1st, 2025. We will enroll as many additional participants as possible until this end-date.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD according to the DSM-5 and related to military service, ages 20-70

Exclusion Criteria:

* Psychotic or Bipolar disorder, drug and alcohol abuse, high risk of harming self or others, other psychological treatment, vision problems that are not overcome with regular glasses, physical disability that prevents ability to operate computer.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Clinician-rated PTSD symptoms from Pre- to Post-Treatment | 1.5-2 months
  Change in total score on the Clinician Administered PTSD Scale (CAPS-5) from pre- to post-treatment
Clinician-rated PTSD symptoms at 3-month Follow-up | 3 Months after treatment completion
  Total score on the Clinician Administered PTSD Scale (CAPS-5) at 3-month Follow-up
Change in PTSD Diagnosis from Pre- to Post-Treatment | 1.5-2 months
  Change in PTSD diagnosis, derived from CAPS-5 corresponding to DSM-5 criteria, from pre- to post-treatment
PTSD Diagnosis at 3-month Follow-up | 3 Months after treatment completion
  PTSD diagnosis derived from CAPS-5 corresponding to DSM-5 criteria at 3-month Follow-up

SECONDARY OUTCOMES:
Change in Patient-rated PTSD symptoms from Pre- to Post-Treatment | 1.5-2 months
  Change in score on self-report questionnaire Posttraumatic stress disorder checklist for DSM-5 (PCL-5) from Pre- to Post-Treatment. The total score, ranging from 0 to 80, reflects PTSD symptom severity, with higher scores representing greater severity.
Patient-rated PTSD symptoms at 3-month Follow-up | 3 Months after treatment completion
  Score on self-report questionnaire Posttraumatic stress disorder checklist for DSM-5 (PCL-5) at 3-month Follow-up. The total score, ranging from 0 to 80, reflects PTSD symptom severity, with higher scores representing greater severity.
Change in Patient-rated Depression symptoms from Pre- to Post-Treatment | 1.5-2 months
  Change in Score on self-report Patient Health Questionnaire 9 (PHQ-9) from Pre- to Post-Treatment. The total score, ranging from 0-27, reflects severity of depressive symptoms, with higher scores representing greater severity.
Patient-rated Depression symptoms at 3-month Follow-up | 3 Months after treatment completion
  Score on self-report Patient Health Questionnaire 9 (PHQ-9) at 3-month Follow-up. The total score, ranging from 0-27, reflects severity of depressive symptoms, with higher scores representing greater severity.
Pre-treatment Clinical Global Impression Scale | Up to 2 weeks pre-treatment
  Clinician Rated Symptom Severity & Improvement. Severity and improvement scales (CGI-S/I) will be used to assess participants global clinical condition. The CGI-S and the CGI-I are single-items, clinician-reported, measure assessing severity and improvement of illness using a 7-point Likert-type scale. The CGI-S/I has good inter-rater reliability and concurrent validity with other measures. This tool is widely used in clinical trials concerning psychopathology treatments and has good sensitivity to clinical change.
Post-treatment Clinical Global Impression Scale | 1-2 weeks post-treatment
  Clinician Rated Symptom Severity & Improvement. Severity and improvement scales (CGI-S/I) will be used to assess participants global clinical condition. The CGI-S and the CGI-I are single-items, clinician-reported, measure assessing severity and improvement of illness using a 7-point Likert-type scale. The CGI-S/I has good inter-rater reliability and concurrent validity with other measures. This tool is widely used in clinical trials concerning psychopathology treatments and has good sensitivity to clinical change.

OTHER OUTCOMES:
Change in behavioral Attention Bias from Baseline to Post-treatment | 1.5-2 months
  Change in Attention Bias will be assessed with two scores, one resulting from a response-time based dotprobe task and another from an eye-tracking computer task.
Behavioral Attention Bias at 3-month Follow-up | 3 Months after treatment completion
  Attention Bias will be assessed again at the 3 month follow-up. It will be measured with two tasks, one response-time based dotprobe task and an eye-tracking computer task.
Change in behavioral Attention Control from Baseline to Post-treatment | 1.5-2 months
  Change in Behavioral Attention Control from Baseline to Post-training Measurement will be assessed using a Flanker computer task.
Behavioral Attention Control at 3-month Follow-up | 3 Months after treatment completion
  Behavioral Attention Control will be assessed again at 3-month Follow-up using a Flanker computer task.
Change in Subjective Attention Bias from Baseline to Post-treatment | 1.5-2 months
  Change in score on self-report Attention Bias Questionnaire (ABQ) from Baseline to Post-treatment. The total score, ranging from 0 to 36, represents threat-related attention bias, with higher scores representing greater bias toward threat.
Subjective Attention Bias at 3-month Follow-up | 3 Months after treatment completion
  Score on subjective Attention Bias Questionnaire (ABQ) at 3-month Follow-up. The total score, ranging from 0 to 36, represents threat-related attention bias, with higher scores representing greater bias toward threat.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lazarov A, Pine DS, Bar-Haim Y. Gaze-Contingent Music Reward Therapy for Social Anxiety Disorder: A Randomized Controlled Trial. Am J Psychiatry. 2017 Jul 1;174(7):649-656. doi: 10.1176/appi.ajp.2016.16080894. Epub 2017 Jan 20. PMID 28103714